CLINICAL TRIAL: NCT06977334
Title: Identification of Ovarian Malignancy With Ultrasonography Based Criteria (IOTA) and Serum CA 125
Brief Title: IOTA Ultrasound Criteria and Serum CA 125 for Ovarian Malignancy Detection
Acronym: IOTA-CA125
Status: Completed | Type: Observational
Sponsor: Maharajgunj Medical Campus (Other)
Responsible Party: Principal Investigator, Amit Yadav, MBBS Doctor, Maharajgunj Medical Campus
Other Study IDs: IRC-NMCTH-08/2021
Record Dates: First submitted 2025-05-09; First posted 2025-05-18 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Ovarian Neoplasms; Ovarian Cancer; Ovarian Carcinoma
Keywords: IOTA; CA 125; Ultrasonography; Ovarian malignancy
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This cross-sectional analytic study assessed the diagnostic accuracy of IOTA Simple Rules versus serum CA 125 in women with adnexal masses undergoing surgery. Eighty-two percent of tumors were classifiable by IOTA criteria; CA 125 cut-offs of 35, 70, and 105 U/mL were evaluated against histopathology gold standard.

DETAILED DESCRIPTION:
All women admitted to the Department of Obstetrics and Gynecology and assigned for the surgery of adnexal mass were enrolled in the study. After written informed consent, the clinical proforma was filled up. Data collection regarding age, current or previous hormonal contraception, menopausal status and family history of breast or ovarian cancer, clinical presentation. Participants were scheduled for ultrasound evaluation done according to IOTA simple rules (five malignant features and five benign features) and peripheral blood was collected for tumor marker serum CA125 measurement.

During ultrasonographic examination, the morphology of the adnexal masses was characterized using 2D real-time and color Doppler ultrasound. Adnexal masses were described according to origin (ovarian/extra ovarian); position (right/left/bilateral); number of lesions; type of lesions (unilocular/unilocular - solid/multilocular/multilocular - solid); size; volume; intracystic fluid echogenicity; number of locations; presence and size of septations; presence, number, size of solid papillary projections; largest solid component; presence / absent of ascites. These parameters are used as designation according to IOTA Group.

For the sample of CA125, approximately 2 ml blood was collected and registered patient's hospital number, then the selected reagent was added to the sample and kept in a fully automated immunoassay system in the hospital laboratory where electrochemiluminescence Immunoassay method (ECLIA) is used for the analysis. Surgery was performed in the hospital and a biopsy was sent for the histopathology examination in the same hospital.

Sensitivity, specificity, positive predictive value, and negative predictive values of CA125 and IOTA class were calculated. The correlation between CA 125 and IOTA simple rules was analyzed and compared with histopathological reports using the Pearson correlation method. The area under the receiver operating characteristic curve (AUC) was used to determine the point at which CA125 had the highest sensitivity and specificity in distinguishing histologically malignant from benign tumors.

ELIGIBILITY:
Inclusion Criteria:

* All age groups and parity with ovarian mass admitted for scheduled surgery.

Exclusion Criteria:

* Proven cases of ovarian malignancy
* Ovarian mass in pregnancy

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: The patient assigned for surgery due to an ovarian tumor in the Department of Obstetrics and Gynecology, Nobel Medical College Teaching Hospital (NOMCTH), Kanchanbari 5, Biratnagar
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Sensitivity of IOTA Simple Rules | At surgery/histopathology
  Proportion of histologically malignant masses correctly identified by IOTA criteria.
Specificity of IOTA Simple Rules | At surgery/histopathology
  Proportion of histologically malignant masses correctly identified by IOTA criteria.
Sensitivity of Serum CA 125 (cut-off 35 U/mL) | Preoperative blood draw
  Proportion of malignant tumors with CA 125 >35 U/mL.
Specificity of Serum CA 125 (cut-off 35 U/mL) | Preoperative blood draw
  Proportion of benign tumors with CA 125 ≤35 U/mL.
Area Under the ROC Curve for CA 125 | Preoperative blood draw vs histopathology
  Discriminatory performance of CA 125 at multiple cut-off points.

CONTACTS AND LOCATIONS:
Overall Officials: Chandrika Dangol, MD, Study Director — Nobel Medical College Teaching Hospital
Locations (1):
- Nobel Medical College Teaching Hospital, Biratnagar, Koshi, Nepal